CLINICAL TRIAL: NCT03711266
Title: Michigan Mental Health Integration Partnership (MIP) - Implementing PTSD Treatment in FQHCs for Michigan Medicaid Enrollees
Brief Title: Implementing PTSD Treatment in FQHCs for Michigan Medicaid Enrollees
Acronym: PE-PC Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Michigan Department of Health and Human Services (Other)
Responsible Party: Principal Investigator, Rebecca Sripada, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00149877
Record Dates: First submitted 2018-10-12; First posted 2018-10-18 (Actual); Results first posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2021-12

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PE-PC (Experimental): Eligible participants who present to participating CHCs and screen positive for PTSD will be offered PE-PC via telepsychiatry.
  Interventions: Behavioral: PE-PC

INTERVENTIONS:
Behavioral: PE-PC — PE-PC treatment will follow the PE-PC manual and patient workbook. Treatment content for PE-PC is drawn from the PE model and condensed so as to deliver the most efficacious components of PE. PE-PC consists of four, 30-minute appointments scheduled approximately once a week over 4-6 weeks

SUMMARY:
The purpose of this project is to expand access to trauma-focused treatment among Medicaid Enrollees with PTSD, thereby improving the quality of mental health services delivered to this population. Specifically, the project goals are to evaluate the delivery and sustainability of a brief trauma-focused treatment, Prolonged Exposure for Primary Care (PE-PC), an evidence-based intervention for PTSD, when delivered via telehealth to patients enrolled at CHCs in Michigan.

DETAILED DESCRIPTION:
This project directly addresses the Michigan Department of Health and Human Services (MDHHS) Mental Health and Wellness commission priority to provide "better access to high quality, coordinated and consistent service and care between agencies, service providers and across geographical boundaries."

The project goals are to evaluate the delivery and sustainability of a brief trauma-focused treatment, Prolonged Exposure for Primary Care (PE-PC), an evidence-based intervention for PTSD, when delivered via telehealth to patients enrolled at CHCs in Michigan. CHCs serve 680,000 Michigan residents across 260 delivery sites. Ninety-two percent of CHC patients have incomes below 200 percent of the federal poverty level. Approximately 16 percent of CHC patients are uninsured, and more than 53 percent rely on Medicaid for their insurance. Thus, providing PTSD treatment to CHC patients will improve care to Medicaid enrollees and promote Mental Health and Wellness commission priorities of developing a trauma informed system that includes implementation of evidence-based trauma-informed care.

To address the high burden of PTSD in Medicaid enrollees in Michigan CHCs, we plan to deliver PE-PC to patients in CHCs. This treatment consists of four 30-minute sessions of in-vivo and narrative exposure, with content drawn from the PE model. Recently published efficacy data from a randomized controlled trial showed that PE-PC significantly reduced PTSD and depression symptoms as compared to usual primary care treatment. These changes were maintained at 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. receive care at a Michigan CHC
2. have a PCL-5 score ≥33
3. have had psychotropic medication stability for at least 4 weeks

Exclusion Criteria:

1. substantially cognitively impaired (according to the Mini-Cog)
2. unable to agree to study procedures for any reason (including incompetency)
3. at high risk of suicide
4. currently engaged in a trauma-focused behavioral treatment (such as Prolonged Exposure or Cognitive Processing Therapy)
5. unable to speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Sripada, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Baldwin Family Health Care-Cadillac Clinic, Cadillac, Michigan
  - Hamilton Community Health Network-Flint Clinic, Flint, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sripada RK, Walters HM, Ganoczy D, Avallone KM, Cigrang JA, Rauch SAM. Feasibility and Acceptability of Prolonged Exposure in Primary Care (PE-PC) for Posttraumatic Stress Disorder in Federally Qualified Health Centers: A Pilot Study. Adm Policy Ment Health. 2022 Sep;49(5):722-734. doi: 10.1007/s10488-022-01195-1. Epub 2022 Apr 20. PMID 35445362

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We aimed to recruit 40-50 patients. However, due to FQHC constraints during the COVID-19 pandemic, we were only able to recruit 35 patients.
Pre-assignment Details: Thirty-five patients were enrolled; however, five were removed by the study therapist prior to intervention initiation and were not included in the final analysis. Three of these patients had a comorbid condition requiring a higher level of care (active psychotic symptoms; severe emotion dysregulation), one was deemed to be at high risk for suicide, and one did not meet diagnostic criteria for PTSD.
Period: Overall Study
Arm/Group | PE-PC
Started | 30
Completed | 20
Not Completed | 10
Not completed — Lost to Follow-up | 10

BASELINE CHARACTERISTICS:
Population: All analyses, including baseline characteristics, were conducted on the 30 enrolled participants, regardless of the number of intervention sessions they attended.
Arm/Group | PE-PC
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (15.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 25
  Male | 4
  Other | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American | 12
  Caucasian | 14
  Multi-racial | 4
  Hispanic or Latino | 4
  Non-Hispanic or Latino | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in PTSD Symptoms (as Measured by the PCL-5)
Description: The PCL-5 is a 20-item self-report measure designed to assess PTSD symptoms as defined by the DSM-5. Each item of the PCL-5 is scored on a five point scale ranging from 0 ("not at all") to 4 ("extremely"). Items are summed to provide a total severity score (range = 0-80).The PCL-5 has strong internal consistency, test-retest reliability, and convergent and discriminant validity. Scores ≥ 33 indicate a probable diagnosis of PTSD. Data presented represent a change from baseline PCL-5 assessment to the 4-month PCL-5 assessment (e.g., value at baseline minus value at 4 months).
Time Frame: Baseline, 4-months
Population: Thirty patients were included in the final analysis. The analysis strategy was intent-to-treat, and multiple imputation was used to impute missing follow-up data. We included auxiliary variables that were correlated with the missing variables at r > 0.4 (Enders, 2010).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PE-PC
Number analyzed (Participants) | 30
score on a scale | 31.4 [18.5 to 44.3]
Statistical Analysis 1: Comparison: PE-PC; Thirty patients were included in the final analysis. The analysis strategy was intent-to-treat, and multiple imputation was used to impute missing follow-up data. We included auxiliary variables that were correlated with the missing variables at r > 0.4 (Enders, 2010); Test type: Other; p < .001, t-test, 2 sided; Mean Difference (Final Values) = 31.4, 95% CI 2-sided [18.5 to 44.3]

2. Secondary Outcome: Change in Depressive Symptoms (as Measured by the PHQ-9)
Description: The PHQ-9 is a 9-item self-report measure that assesses the presence and severity of depressive symptoms. Patients are asked to rate the presence of symptoms over the past 2 weeks on a 4-point likert scale ranging from 0-3 (not at all, several days, more than half the days, nearly every day) with a range of scores between 0-27. Total scores ranging from 5-9 indicate mild depression, 10-14 indicate moderate depression, 15-19 indicate moderately severe depression, and 20-27 indicate severe depression. Data presented represent a change from baseline PHQ-9 assessment to the 4-month PHQ-9 assessment (e.g., value at baseline minus value at 4 months).
Time Frame: Baseline, 4-months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | PE-PC
Number analyzed (Participants) | 30
score on a scale | 8.5 [3.7 to 13.3]

3. Secondary Outcome: Change in Recovery Goals (Measured by the Recovery Assessment Scale; RAS)
Description: Recovery orientation will be measured using the Recovery Assessment Scale - Short Form (RAS-SF). This 20-item scale is a shorter version of the RAS and has four factors: personal confidence and hope, willingness to ask for help, reliance on others, and no domination by symptoms. All items on the RAS assessment are rated on a 5-point Likert scale: 1 = Strongly Disagree, 2 = Disagree, 3 = Not Sure, 4 = Agree, and 5 = Strongly Agree with a range of scores between 20-100. All items are summed to compute a total score. Higher scores indicate greater recovery orientation. The RAS-SF shows evidence for both convergent and discriminant validity when compared to quality of life, social support, and symptomatic scales. Data presented represent a change from baseline RAS-SF assessment to the 4-month RAS-SF assessment (e.g., value at baseline minus value at 4 months)).
Time Frame: Baseline, 4-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PE-PC
Number analyzed (Participants) | 30
score on a scale | 9.57 (16.34)

4. Secondary Outcome: Change in Posttraumatic Cognitions (Measured by the Post-Traumatic Cognitions Inventory; PTCI)
Description: The PTCI is a 33-item scale of trauma-related thoughts and beliefs which is rated on a Likert-type scale ranging from 1 (totally disagree) to 7 (totally agree). It is composed of 3 subscales. Each subscale is calculated by averaging the items in the subscale. The PTCI total score is calculated as the sum of the three subscales and ranges from 3 to 21. Results reported here are total scores, not subscale scores. Higher scores represent more dysfunctional cognitions. Data presented represent a change from baseline PTCI assessment to the 4-month PTCI assessment (e.g., value at baseline minus value at 4 months).
Time Frame: Baseline, 4-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PE-PC
Number analyzed (Participants) | 30
score on a scale | 2.65 (4.04)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the period of time the participants were enrolled in the study. For this study, that period of time included 8 months.
Description: The study followed standard AE/SAE reporting guidelines.
Arm/Group | PE-PC
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT03711266/Prot_SAP_000.pdf